CLINICAL TRIAL: NCT02116270
Title: Accelerated Immunosenescence and Chronic Kidney Disease
Acronym: IRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRIS API/2012/28
Record Dates: First submitted 2014-04-09; First posted 2014-04-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-08

CONDITIONS: Renal Failure
Keywords: Renal Failure; Dialysis; Biological Aging
MeSH Terms: conditions — Renal Insufficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (Other): Patients in this group control (normal renal function) are followed in the urology department. A blood sample is performed on the day of inclusion.
  Interventions: Biological: Blood sample
- Severe renal failure (Experimental): Patients in this group suffer from renal failure stage 4 and are not under dialysis. A blood sample is performed on the day of inclusion.
  Interventions: Biological: Blood sample
- Peritoneal dialysis (Experimental): Patients with renal failure, under peritoneal dialysis for at least 3 months. A blood sample is performed on the day of inclusion.
  Interventions: Biological: Blood sample
- Hemodialysis (Experimental): Patient with renal failure, under hemodialysis for at least 3 months. A blood sample is performed on the day of inclusion.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — 3 tubes of 5 ml tubes and 4 of 7 ml for biological assays at t0.

SUMMARY:
The aim of this study is to investigate the impact of renal function and dialysis techniques on the percentage of senescent T lymphocytes.

DETAILED DESCRIPTION:
The immunosenescence is a complex and profound remodeling of the immune system during life. It is mainly due to thymic involution and repeated antigenic stimulation. Kidney disease is associated with a decrease in adaptive immunity as evidenced by the decrease in vaccine response and increased susceptibility to infections, similar to those observed in the elderly population.

However, data on aging of the immune system in chronic kidney disease remains incomplete. Furthermore, the determinants of immunosenescence are not also not known. It is possible that "uremic" factors help explain the phenotypic and functional changes of lymphocytes, as antigenic stimuli associated with repeated bio-compatible materials used in dialysis contact.

The purpose of this study is to describe the phenotypes of the immune system of renal and analyze the determinants of these changes.

ELIGIBILITY:
Inclusion Criteria:

* Patient able to understand the reason of the study
* Patient not opposed to the conservation of biological samples for scientific research

Exclusion Criteria:

* Patient suffering from psychotic illness
* Any history of immunosuppressive therapy (except steroids up to 5mg/day)
* History of cancer (except skin cancer) or treated hematological malignancy
* Infectious episode required hospitalization not older 3 months
* Hepatitis B or C infection
* HIV infection, active or inactive
* For dialysis patients: renal failure on dialysis for less than 3 months and/or have benefited from two techniques for renal replacement therapy in the last 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Cluster of Differentiation (CD) 4/8+ CD 57+ CD 28- lymphocytes (senescent lymphocytes) | 6 months
  The primary outcome measure is the percentage of CD 4/8+ CD 57+ CD 28- lymphocytes by flow cytometry. The technique used is a 6 colors surface labelling of T lymphocytes to study the T cell senescent population.

SECONDARY OUTCOMES:
Telomerase Activity of T lymphocytes | 6 months
  The telomerase activity of T lymphocytes is assessed by a method of Polymerase chain reaction (PCR)-ELISA.
Level of phospho-histone 2AX (gH2AX) in peripheral blood T lymphocytes | 6 months
  This level is obtained by flow cytometry after permeabilization and labelling of Peripheral Blood Mononuclear Cells (PBMC).
Proportion of Recent Thymic Emigrants (RTE) in peripheral blood T lymphocytes | 6 months
  RTE T cells will be defined by flow cytometry, according to co-expression of CD 4, CD 8,CD 31 and CD 45RA
T-cell receptor excision circle (TREC) level in PBMC. | 6 months
  TRECs study is based on a technique of quantitative PCR using DNA extracted from PBMC.
Telomere length in T lymphocytes | 6 months
  Study of telomere length is performed after extraction of DNA from isolated T cells. The length is determined by a quantitative PCR technique relative to a reference gene.

CONTACTS AND LOCATIONS:
Overall Officials: Jamal BAMOULID, Doctor, Principal Investigator — CHU de Besançon
Locations (1):
- Service de néphrologie, CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No